CLINICAL TRIAL: NCT01474954
Title: A Phase 2b Randomized, Double-Blind, Double-Dummy Trial of 100 or 200 mg Once-Daily Doses of Cenicriviroc (CVC, TBR-652) or Once-Daily EFV, Each With Open-Label FTC/TDF, in HIV-1-Infected, Antiretroviral Treatment-Naïve, Adult Patients With Only CCR5-Tropic Virus
Brief Title: Investigation of The Effect of Cenicriviroc (CVC) Plus FTC/TDF on Cardiovascular Disease Risk Factors
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 652-2-202
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infection
Keywords: HIV; Antiretroviral Medication; Cardiovascular Disease Risk
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a single-site substudy, "Investigation of the Effect of Cenicriviroc (CVC) plus Emtricitabine/Tenofovir (FTC/TDF) on Atherosclerosis Risk Factors", open to all patients enrolled in the primary study, "A Phase 2b Randomized, Double-Blind, Double-Dummy Trial of 100 or 200 mg Once-Daily Doses of Cenicriviroc (CVC, TBR-652) or Once-Daily EFV, Each With Open-Label FTC/TDF, in HIV-1-Infected, Antiretroviral Treatment-Naïve, Adult Patients With Only CCR5-Tropic Virus", in the San Francisco Bay area to evaluate changes in brachial flow mediated dilation in patients in one of three treatment groups: 1. Cenicriviroc (CVC) at 100mg (2 tablets, 50mg each) QD + CVC matching placebo (2 tablets) QD + Efavirenz (EFV) matching placebo (1 capsule) QHS + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (1 tablet) QD; 2. CVC at 200mg (4 tablets, 50mg each) QD + EFV matching placebo (1 capsule) QHS + FTC/TDF (1 tablet) QD; 3. CVC matching placebo (4 tablets) QD + EFV 600 mg (1 capsule) QHS + FTC/TDF (1 tablet) QD. The substudy will run for the duration of the primary study. 50 patients of the 150 total enrolled in the primary study will be referred to and enrolled in the cardiovascular substudy.

Patients enrolled in the substudy and substudy protocol staff will be blinded to study treatment. Data obtained on this substudy will be analyzed in conjunction with laboratory data for cardiovascular disease risk factors and HIV-1 RNA levels obtained on the primary study.

The primary study is a randomized, double-blind, double-dummy, 48-week, comparative study in approximately 150 HIV-1-infected, treatment-naïve patients with CCR5-tropic virus. Patients will be stratified by Screening HIV-1 RNA level (≥100,000 copies/mL versus <100,000 copies/mL) and randomized 2:2:1 to one of the three treatment groups. Patients will receive all medications from the primary study, and thus the primary study site will be responsible for any adverse outcomes with the drug.

DETAILED DESCRIPTION:
This is a single-site substudy, "Investigation of the Effect of Cenicriviroc (CVC) plus Emtricitabine/Tenofovir (FTC/TDF) on Atherosclerosis Risk Factors", open to all patients enrolled in the primary study, "A Phase 2b Randomized, Double-Blind, Double-Dummy Trial of 100 or 200 mg Once-Daily Doses of Cenicriviroc (CVC, TBR-652) or Once-Daily EFV, Each With Open-Label FTC/TDF, in HIV-1-Infected, Antiretroviral Treatment-Naïve, Adult Patients With Only CCR5-Tropic Virus", in the San Francisco Bay area to evaluate changes in brachial flow mediated dilation in patients in one of three treatment groups: 1. Cenicriviroc (CVC) at 100mg (2 tablets, 50mg each) QD + CVC matching placebo (2 tablets) QD + Efavirenz (EFV) matching placebo (1 capsule) QHS + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (1 tablet) QD; 2. CVC at 200mg (4 tablets, 50mg each) QD + EFV matching placebo (1 capsule) QHS + FTC/TDF (1 tablet) QD; 3. CVC matching placebo (4 tablets) QD + EFV 600 mg (1 capsule) QHS + FTC/TDF (1 tablet) QD. The substudy will run for the duration of the primary study. 50 patients of the 150 total enrolled in the primary study will be referred to and enrolled in the cardiovascular substudy.

Patients enrolled in the substudy and substudy protocol staff will be blinded to study treatment. Data obtained on this substudy will be analyzed in conjunction with laboratory data for cardiovascular disease risk factors and HIV-1 RNA levels obtained on the primary study.

The primary study is a randomized, double-blind, double-dummy, 48-week, comparative study in approximately 150 HIV-1-infected, treatment-naïve patients with CCR5-tropic virus. Patients will be stratified by Screening HIV-1 RNA level (≥100,000 copies/mL versus <100,000 copies/mL) and randomized 2:2:1 to one of the three treatment groups. Patients will receive all medications from the primary study, and thus the primary study site will be responsible for any adverse outcomes with the drug.

Primary Objective:

· To assess changes from Baseline in brachial artery vascular patency after 24 weeks of treatment with a CVC containing regimen.

Secondary Objectives:

* To compare changes from Baseline in vascular patency and after 48 weeks of treatment with CVC versus EFV.
* To assess changes from Baseline to Weeks 4, 12, 24, and final follow-up in vascular patency.
* To assess changes from Baseline to Week 48 in flow-mediated dilation (FMD) in relation to immunologic and metabolic covariates.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female, HIV-1-infected patients 18 years old and older.
* Body mass index (BMI) 18 to <=35 kg/m2
* Antiretroviral treatment-naive (no prior non-nucleoside reverse transcriptase inhibitor, other than in women who received a single dose of perinatal nevirapine who have no K103 viral mutation, no prior CCR5 antagonist therapy, no more than 10 days of any other prior antiretroviral therapy)
* HIV-1 CCR5-tropic-only virus, as determined on both a tropism genotype and the enhanced Trofile assay
* Plasma HIV-1 RNA level >= 1,000 copies/mL at Screening Visit 1
* CD4 count >= 250 cells/mm3 at Screening Visit 1
* Able and willing to provide written informed consent
* Willing to take appropriate precautions to prevent pregnancy
* Women of child-bearing potential may be enrolled following a negative urine pregnancy test. If participating in activity that could lead to pregnancy, men and women must agree to use two forms of barrier method contraception during the trial and for 3 months after stopping the medication.
* Women who are not of reproductive potential (documented to be surgically sterile or postmenopausal [defined as amenorrhea >= 1 year and follicle stimulating hormone>= 30 mU/mL]) are eligible to be enrolled
* Signed informed consent for participation in the sub-study

Exclusion Criteria:

* Presence of CXCR4- or dual/mixed-tropic HIV-1 virus on either the enhanced Trofile assay or a tropism genotype
* Presence of primary resistance mutations or phenotypic resistance to TDF, FTC, or EFV and/or mutations associated with multidrug nucleoside/nucleoside resistance
* An active CDC category C disease (except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial)
* Any historical CD4 count <200 cells/mm3
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value Grade >=2 or total bilirubin greater than the upper limit of normal (ULN) during Screening
* History of HIV-2, hepatitis B and/or C, cirrhosis of the liver, or any known active or chronic liver disease. Hepatitis B vaccinated patients are eligible, as follows:
* Patients with a recent history of hepatitis B (positive hepatitis B surface antigen [HBsAg]) are excluded.
* Patients with prior exposure to hepatitis B but with no virus present (positive hepatits B surface antibody [HBsAb]) are eligible provided liver function tests (AST and ALT) are within normal ranges, the patient has no signs/symptoms of hepatitis, and all other entry criteria are met.
* Patients with positive hepatitis B core antibody (HBcAb) may be chronic carriers of hepatitis B or have cleared the virus and are eligible provided liver function tests (AST and ALT) are completely normal, the patient has no signs/symptoms of hepatitis, and all other entry criteria are met.
* Patients with positive hepatitis C antibody (HCVAb) are excluded, except those with proof of viral clearance and normal liver function tests (LFTs) may be eligible with Medical Monitor approval.
* A current diagnosis of tuberculosis (TB) infection, any prior untreated TB infection, inadequate treatment of active TB, or inadequate treatment for a positive purified protein derivative (PPD) test. Cases of active infection and latent TB infection with a documented history of adequate treatment may be considered for enrollment provided the subject has a negative chest x-ray following treatment and within 6 months before randomization. Adequate treatment is defined as meeting the current recommendations of the Centers for Disease Control and Prevention (CDC). National Institutes of Health (NIH), and the HIV Medicine Association of the Infectious Diseases Society of America (IDSA) guidelines, or other CDC recommendations if the patient was treated before the current recommendations or before coinfection with HIV. Investigators are encouraged to discuss such cases with the Medical Monitor if in doubt as to patient eligibility.
* Any prior or current diagnosis with other intracellular pathogens.
* Recent history (<30 days) of clinically significant infection or illness.
* Pregnancy or breastfeeding
* Current or anticipated treatment with immunmodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity
* Immunization within 30 days of first dose of investigational study drug.
* Current alcohol or durg use, which in the expert judgment of the Investigator, will interfere with the patient's ability to comply with the protocol requirements.
* Any experimental medication within 30 days prior to Screening or anticipated use during the trial.
* Current (within 5 half-lives or 14 days prior to the first dose of study drug, whichever is longer) or anticipated use of antimetabolites; alkylating agents; or drugs, herbal preparations (including St. John's wort), and foods (including grapefruit) known to affect the cytochrom P450 (CYP) family CYP 3A4 or CYP 2C8 enzymes or P-glycoprotein (P-gp) transporters.
* Use of over-the counter (OTC) medications as follows:
* In the first 25 patients, any systemic OTC preparations, including herbal preparations (e.g. phytotherapeutic, herbal, or plant-derived preparations), within 14 days prior to the first dose of study medication)
* After the first 25 patients, systemic OTC herbal medications (including phytotherapeutic, herbal, or plant-derived preparations) within 14 days prior to the first dose of study medication, unless approved by the Investigator.
* After the first 25 patients, chronically needed OTC medications, unless discussed with and approved by the Medical Monitor
* History of clinically significant metabolic, endocrine, hepatic, renal, hematologic, pulmonary, gastrointestinal, or cardiovascular disorders.
* Uncontrolled hypertension (i.e. systolic blood pressure [BP] >=140 or diastolic BP >= 90)
* Bradycardia, defined as sinus rhythm <50 beats/min (bpm)
* History or presence of an abnormal electrocardiogram (ECG)
* Presence of any condition that would interfere with the absorption, distribution, metabolism, or excretion of the drug.
* After the first 25 patients enrolled, adequately controlled conditions such as gastroesophageal reflux disease (GERD) may be allowed. Investigators are encouraged to discuss such cases with the Medical Monitor if in doubt as to patient eligibility.
* History of malignancy except cured basal or squamous cell carcinoma of the skin
* Patients who have received radiation or cytotoxic chemotherapeutic agents, unless fully recovered by the time of the first dose of study drug, or who may require them during the study period.
* Patients who are, in the opinion of the Investigator, unable to comply with the dosing schedule and protocol evaluations.
* Inability to access the research clinic.
* Inability, in the judgement of the investigator, to comply with the additional requirements of the sub-study.
* Starting, stopping, or changing lipid-lowering antihypertensive medications within the 12 weeks before study entry.
* Persistent resting blood pressure of less than 100/70 mm Hg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All primary study participants who received at least one dose of study drug and had data from both a Baseline and at least 1 post-Baseline vis.t
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess changes from Baseline in brachial artery vascular patency after 24 weeks of treatment with a CVC containing regimen. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — San Francisco General Hospital
Locations (1):
- University of California, San Francisco; San Francisco General Hospital, San Francisco, California, United States